CLINICAL TRIAL: NCT03556969
Title: Use of Perfusion Index Change as a Predictor of Hypotension During Propofol Sedation in Adult Patients Undergoing Hip Surgery Under Spinal Anesthesia: A Prospective Observational Study
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hwan Lee, Associate Professor, Samsung Medical Center
Other Study IDs: 2018-03-052
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Hypotension; Spinal Anesthetics Causing Adverse Effects in Therapeutic Use
MeSH Terms: conditions — Hypotension | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Propofol sedation after SA: Participants who undergo propofol sedation after spinal anesthesia
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — no intervention

SUMMARY:
This observational study is to evaluate Perfusion Index Change as a Predictor of Hypotension During Propofol Sedation in Adult Patients Undergoing Hip Surgery Under Spinal Anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients having hip surgery under spinal anesthesia and propofol sedation

Exclusion Criteria:

* ASA class IV or above
* pregnancy
* inability to measure noninvasive blood pressure on the arm
* preexisting hemodynamic instability
* known peripheral artery occlusive disease
* known autonomic nerve dysfunction
* uncontrolled hypertension

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from both genders, ranging from young to very old patients.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
5-minute perfusion index change | After sedation until start of surgery (an average of 20 minutes)
  ability of perfusion index change 5 minutes after induction in predicting propofol sedation-induced hypotension (perfusion index change is calculated as the percent change from baseline values)
10-minute perfusion index change | After sedation until start of surgery (an average of 20 minutes)
  ability of perfusion index change 10 minutes after induction in predicting propofol sedation-induced hypotension (perfusion index change is calculated as the percent change from baseline values)
baseline perfusion index | After sedation until start of surgery (an average of 20 minutes)
  ability of baseline perfusion index in predicting propofol sedation-induced hypotension
5-minute perfusion index | After sedation until start of surgery (an average of 20 minutes)
  ability of perfusion index 5 minutes after induction in predicting propofol sedation-induced hypotension
10-minute perfusion index | After sedation until start of surgery (an average of 20 minutes)
  ability of perfusion index 10 minutes after induction in predicting propofol sedation-induced hypotension

SECONDARY OUTCOMES:
5-minute perfusion index change difference | After sedation until start of surgery (an average of 20 minutes)
  difference of perfusion index change 5 minutes after induction between participants who do or do not develop hypotension during propofol sedation after spinal anesthesia (perfusion index change is calculated as the percent change from baseline values)
10-minute perfusion index change difference | After sedation until start of surgery (an average of 20 minutes)
  difference of perfusion index change 10 minutes after induction between participants who do or do not develop hypotension during propofol sedation after spinal anesthesia (perfusion index change is calculated as the percent change from baseline values)
baseline perfusion index difference | After sedation until start of surgery (an average of 20 minutes)
  difference of baseline perfusion index between participants who do or do not develop hypotension during propofol sedation after spinal anesthesia
5-minute perfusion index difference | After sedation until start of surgery (an average of 20 minutes)
  difference of perfusion index after 5 minutes of induction between participants who do or do not develop hypotension during propofol sedation after spinal anesthesia
10-minute perfusion index difference | After sedation until start of surgery (an average of 20 minutes)
  difference of perfusion index after 10 minutes of induction between participants who do or do not develop hypotension during propofol sedation after spinal anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Sungkyunkwan University, School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided